CLINICAL TRIAL: NCT00627237
Title: Short-Term Executive Plus (STEP): A Randomized Controlled Trial of Short Term Intensive Cognitive Rehabilitation.
Brief Title: Improving Executive Functioning After Traumatic Brain Injury (TBI): A Trial of the "Short Term Executive Plus" Program
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GCO 06-0939; CE001171
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injuries; Cognitive Rehabilitation; Executive Functioning
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate start (Experimental): Starts the 12 week intervention immediately after enrollment
  Interventions: Behavioral: Immediate Start
- Waitlist group (Experimental): Starts the 12 week intervention 12 weeks after initial enrollment
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Immediate Start — Participation in an intensive cognitive rehabilitation program 3 days a week (3 hours a day) for 12 weeks. Each day consists of a 50 minutes of problem solving group, 50 minutes of individualized attention training, and a 50 minute emotional regulation group session with 10 minutes breaks between each module.
  Arms: Immediate start
Behavioral: Waitlist — Participation in an intensive cognitive rehabilitation program 3 days a week (3 hours a day) for 12 weeks. Each day consists of a 50 minutes of problem solving group, 50 minutes of individualized attention training, and a 50 minute emotional regulation group session with 10 minutes breaks between each module.
  Arms: Waitlist group

SUMMARY:
The purpose of this study is to determine the efficacy of an intensive short term cognitive rehabilitation program aimed towards improving executive functioning in individuals with traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Executive dysfunction following brain injury (BI) is commonly observed and has been well documented in the literature (Mateer, 1999; Prigatano, 1999; Levine et al., 2000; Shallice & Burgess, 1991; Cicerone & Giacino, 1992; Goldman-Rakic, 1993; Lezak, 1995, Riegal & Gauggel, 2002; McDonald, 2002; Stuss and Levine, 2003). Level of functioning such as vocational success, community reintegration, and social autonomy are associated with executive functioning abilities following BI (Mazaux et al. 1997, Sohlberg, Mateer, & Stuss, 1993; (Stuss & Levine, 2002, McDonald, 2002). Studies describing the rehabilitation of executive dysfunction have been limited to mostly single case or small group designs (Cicerone, et al., 2000). However, there have been three small randomized clinical trials that have had promising results suggesting the need for more research in this area. When considering all of the studies, it is evident that emphasis has been placed on three areas of intervention: attention remediation, emotional regulation and problem-solving. Consequently, given the pervasive disability found in individuals with BI that is secondary to executive function disorders and the promising, but limited, success of problem-solving-based interventions for executive functions, a randomized controlled trial (RCT) of the efficacy of a short-term, intensive executive function training program (Short-Term Executive Plus) is proposed. The Short-Term Executive Plus (STEP) program will combine treatments and treatment approaches that have proved to be effective in previous studies and will be compared to "wait-list" control group. This design was chosen because no appropriate control intervention exists. In other words there is no "standard" rehabilitation treatment available to these individuals that could serve as an appropriate "control" condition/treatment. As discussed earlier, cognitive remediation is typically delivered in extended full-time day treatment programs or weekly/bi-weekly individual sessions. Using more traditional extended treatments as a control condition would be inappropriate, as persons who can participate in extended, full-time are not the target of the proposed intervention. It is hypothesized that the STEP program will result in significant improvements in executive functioning (and related areas of attention, memory, community participation, and life satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old or older;
* Having a TBI as a result of a blow to the head followed by a loss of consciousness or period of being dazed and confused or a period of post traumatic amnesia or clinical signs of altered neurological function; this information must be medically documented (e.g., emergency medical record, hospital record, neuroradiological report, or neurological exam or record of physician's visit within 24 hours of injury);
* Being at least three months post-injury;
* Being English-speaking (treatment sessions will be conducted in English);
* Reporting executive dysfunction (by self or family);
* Being willing and able to participate in and travel to the program daily for three months;
* Being oriented to time, place and person;
* Having a full-scale IQ of at least 75;
* Having a score on the Galveston Orientation and Amnesia Test of 75 or more;
* Having communication skills adequate to participate in groups;
* Having at least a sixth-grade reading level (for testing and use of written materials);
* Being willing to complete questionnaires and interviews about mood, thinking skills, participation and the like; AND
* Agreeing to participate, i.e., completion of informed consent and HIPAA documents.

Exclusion Criteria:

* Have diminished mental capacity and as a result, are unable to sign informed consent;
* Active substance abuse;
* Active psychosis;
* Active suicidality;
* Disruptive or violent behavior to self or others;
* Current cognitive rehabilitation (this will not include current psychotherapy);
* No impairment on the FRSBE or WCST; OR
* Showing evidence of or a diagnosis of dementia or mild cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Executive functioning | At the beginning of the intervention
Executive functioning | At 12 weeks
Executive functioning | At 24 weeks
Executive functioning | At 6 months
Executive functioning | At 1 year post-intervention.

SECONDARY OUTCOMES:
Attention | At the beginning of the intervention
Attention | At 12 weeks
Attention | At 24 weeks
Attention | At 6 months
Attention | At 1 year post-intervention
Depression and anxiety | At the beginning of the intervention
Depression and anxiety | At 12 weeks
Depression and anxiety | At 24 weeks
Depression and anxiety | At 6 months
Depression and anxiety | At 1 year post-intervention
Memory and learning | At the beginning of the intervention
Memory and learning | At 12 weeks
Memory and learning | At 24 weeks
Memory and learning | At 6 months
Memory and learning | At 1 year post-intervention
Participation, life satisfaction, and self-efficacy | At the beginning of the intervention
Participation, life satisfaction, and self-efficacy | At 12 weeks
Participation, life satisfaction, and self-efficacy | At 24 weeks
Participation, life satisfaction, and self-efficacy | At 6 months
Participation, life satisfaction, and self-efficacy | At 1 year post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Gordon, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Cantor J, Ashman T, Dams-O'Connor K, Dijkers MP, Gordon W, Spielman L, Tsaousides T, Allen H, Nguyen M, Oswald J. Evaluation of the short-term executive plus intervention for executive dysfunction after traumatic brain injury: a randomized controlled trial with minimization. Arch Phys Med Rehabil. 2014 Jan;95(1):1-9.e3. doi: 10.1016/j.apmr.2013.08.005. Epub 2013 Aug 27. PMID 23988395